CLINICAL TRIAL: NCT04879628
Title: A Phase 2, Double-blind, Randomized, Placebo-controlled Study Assessing Efficacy and Safety of SAR441344, a CD40L-antagonist Monoclonal Antibody, in Participants With Relapsing Multiple Sclerosis
Brief Title: Proof-of-concept Study for SAR441344 (Frexalimab) in Relapsing Multiple Sclerosis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACT16877; U1111-1260-3962 (Registry Identifier: ICTRP); 2024-513527-17-00 (Registry Identifier: CTIS); 2020-004785-19 (EudraCT Number)
Record Dates: First submitted 2021-05-06; First posted 2021-05-10 (Actual); Results first posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-08

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Part A is a 12-week, double-blind, placebo-controlled part; Part B is an open-label SAR441344 treatment part.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Intravenous (IV) SAR441344 (Experimental): SAR441344 IV
  Interventions: Drug: SAR441344 IV; Drug: MRI contrast-enhancing preparations
- IV Placebo (Placebo Comparator): Placebo IV
  Interventions: Drug: placebo IV; Drug: MRI contrast-enhancing preparations
- Subcutaneous (SC) SAR441344 (Experimental): SAR441344 SC
  Interventions: Drug: SAR441344 SC; Drug: MRI contrast-enhancing preparations
- SC Placebo (Placebo Comparator): Placebo SC
  Interventions: Drug: placebo SC; Drug: MRI contrast-enhancing preparations

INTERVENTIONS:
Drug: SAR441344 IV — Pharmaceutical form: Solution Route of administration: IV infusion
  Arms: Intravenous (IV) SAR441344
Drug: placebo IV — Pharmaceutical form: Solution Route of administration: IV infusion
  Arms: IV Placebo
Drug: SAR441344 SC — Pharmaceutical form: Solution Route of administration: SC injection
  Arms: Subcutaneous (SC) SAR441344
Drug: placebo SC — Pharmaceutical form: Solution Route of administration: SC injection
  Arms: SC Placebo
Drug: MRI contrast-enhancing preparations — gadolinium compound, including but not limited to Magnevist, Multihance, Prohance, or Elucirem

SUMMARY:
Primary Objective:

To determine the efficacy of SAR441344 as measured by reduction of the number of new active brain lesions

Secondary Objective:

* To evaluate efficacy of SAR441344 on disease activity as assessed by other MRI measures
* To evaluate the safety and tolerability of SAR441344
* To evaluate pharmacokinetics of SAR441344

DETAILED DESCRIPTION:
The duration of each participant will be no longer than 320weeks in both parts of the study, including 4 weeks of screening, at maximum 292 weeks of treatment and 24 weeks of follow-up.

ELIGIBILITY:
Inclusion criteria:

* Participant must be 18 to 55 years of age inclusive, at the time of signing the informed consent.
* The participant must have been diagnosed with RMS (relapsing-remitting MS and secondary progressive MS participants with relapses) according to the 2017 revision of the McDonald diagnostic criteria.
* The participant must have at least 1 documented relapse within the previous year, or ≥2 documented relapses within the previous 2 years, or ≥1 active Gd-enhancing brain lesion on an MRI scan in the past 6 months and prior to screening.
* Body weight within 45 to 120 kg (inclusive) and body mass index (BMI) within the range 18.0 to 35.0 kg/m2 (inclusive) at Screening.
* Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Capable of giving signed informed consent.

Exclusion criteria:

* The participant was diagnosed with PPMS according to the 2017 revision of the McDonald diagnostic criteria or with non-relapsing SPMS.
* The participant had conditions or situations that would adversely affect participation in this study.
* The participant had a history of or currently has concomitant medical or clinical conditions that would adversely affect participation in this study.
* History, clinical evidence, suspicion or significant risk for thromboembolic events, as well as myocardial infarction, stroke and/or antiphosholipid syndrome and any participants requiring antithrombotic treatment.
* Allergies to humanized monoclonal antibodies or severe post-treatment hypersensitivity reactions other than localized injection site reaction, to any biological molecule.
* The participant had received any of the forbidden medications/treatments within the specified time frame before any baseline assessment.
* The participant had taken other investigational drug within 3 months or 5-half-live, whichever is longer, before the screening visit.
* The participant had an EDSS score >5.5 at the first screening visit.
* The participant had a relapse in the 30 days prior to randomization.
* Positive human immunodeficiency virus (HIV) serology (anti HIV1 and anti HIV2 antibodies) or a known history of HIV infection, active or in remission.
* Abnormal laboratory test(s) at Screening.
* Presence of Hepatitis B surface antigen (HBsAg) or anti-Hepatitis B core antibodies (anti-HBc Ab) at screening or within 3 months prior to first dose of study intervention.
* Positive Hepatitis C antibody test result at screening or within 3 months prior to starting study intervention.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 129 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2022-09-21 (Actual); Study Completion 2027-08-23 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (37):
- United States (4):
  - Center for Neurology and Spine- Site Number : 8400007, Phoenix, Arizona
  - University of South Florida Site Number : 8400001, Tampa, Florida
  - The Neurological Institute Site Number : 8400004, Charlotte, North Carolina
  - Medical College of Wisconsin- Site Number : 8400006, Milwaukee, Wisconsin
- Bulgaria (3):
  - Investigational Site Number : 1000002, Pleven
  - Investigational Site Number : 1000003, Sofia
  - Investigational Site Number : 1000001, Sofia
- Investigational Site Number : 1240001, Gatineau, Quebec, Canada
- Czechia (5):
  - Investigational Site Number : 2030003, Brno
  - Investigational Site Number : 2030002, Hradec Králové
  - Investigational Site Number : 2030001, Jihlava
  - Investigational Site Number : 2030005, Ostrava - Poruba
  - Investigational Site Number : 2030004, Teplice
- Investigational Site Number : 2500006, Calais, France
- Germany (2):
  - Investigational Site Number : 2760012, Leipzig
  - Investigational Site Number : 2760004, Münster
- Russia (8):
  - Investigational Site Number : 6430002, Kazan'
  - Investigational Site Number : 6430007, Moscow
  - Investigational Site Number : 6430006, Moscow
  - Investigational Site Number : 6430001, Moscow
  - Investigational Site Number : 6430003, Saint Petersburg
  - Investigational Site Number : 6430005, Saint Petersburg
  - Investigational Site Number : 6430004, Saint Petersburg
  - Investigational Site Number : 6430008, Tyumen
- Spain (2):
  - Investigational Site Number : 7240004, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240002, Vigo
- Turkey (Türkiye) (4):
  - Investigational Site Number : 7920004, Eskişehir
  - Investigational Site Number : 7920003, Istanbul
  - Investigational Site Number : 7920001, İzmit
  - Investigational Site Number : 7920002, Mersin
- Ukraine (7):
  - Investigational Site Number : 8040010, Dnipro
  - Investigational Site Number : 8040006, Dnipro
  - Investigational Site Number : 8040008, Ivano-Frankivsk
  - Investigational Site Number : 8040002, Kyiv
  - Investigational Site Number : 8040004, Lviv
  - Investigational Site Number : 8040003, Odesa
  - Investigational Site Number : 8040005, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Vermersch P, Granziera C, Mao-Draayer Y, Cutter G, Kalbus O, Staikov I, Dufek M, Saubadu S, Bejuit R, Truffinet P, Djukic B, Wallstroem E, Giovannoni G; Frexalimab Phase 2 Trial Group. Inhibition of CD40L with Frexalimab in Multiple Sclerosis. N Engl J Med. 2024 Feb 15;390(7):589-600. doi: 10.1056/NEJMoa2309439. PMID 38354138

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 38 centers in 10 countries. A total of 176 participants were screened from 07 June 2021 to 08 June 2022, of which 47 were screen failures. Screen failures were mainly due to not meeting the eligibility criteria. Primary results are presented up to primary completion date (PCD) of 21 September 2022.
Pre-assignment Details: A total of 129 participants were randomized in a 4:4:1:1 ratio to receive either intravenous (IV) SAR441344 or subcutaneous (SC) SAR441344 or IV placebo or SC placebo in Part A (double-blind [DB] period). After completing Part A, all participants entered Part B (open-label extension [OLE] period) where participants in the IV and SC placebo arms switched to corresponding IV and SC SAR441344 arms and participants from SAR441344 arms continued their previous IV or SC treatment after Week 12 visit.
Groups:
- SC Placebo: Participants received placebo matched to SAR441344 IV infusion loading dose on Day 1 followed by placebo matched to SAR441344 SC injection on Weeks 2, 4, 6, 8 and 10 in Part A (DB period). At Week 12, all participants from this arm switched to active SC SAR441344 300 milligram (mg) every 2 weeks (q2w) and then switched to high SC SAR441344 dose of 1800 mg every 4 weeks (q4w) in Part B (OLE period).
- IV Placebo: Participants received placebo matched to SAR441344 loading dose on Day 1 followed by placebo matched to SAR441344 IV infusion at Weeks 4 and 8 in Part A (DB period). At Week 12, all participants from this arm switched to active IV SAR441344 1200 mg infusion q4w in Part B (OLE period).
- SC SAR441344 300 mg: Participants received SAR441344 600 mg IV infusion loading dose on Day 1 followed by SAR441344 300 mg SC injection on Weeks 2, 4, 6, 8 and 10 in Part A (DB period). At Week 12, participants continued to receive SAR441344 300 mg SC injection q2w and then switched to high SC SAR441344 dose of 1800 mg q4w in Part B (OLE period).
- IV SAR441344 1200 mg: Participants received SAR441344 1800 mg loading dose on Day 1 followed by SAR441344 1200 mg IV infusion at Weeks 4 and 8 in Part A (DB period). At Week 12, participants continued to receive SAR441344 1200 mg IV infusion q4w in Part B (OLE period).
Period: Part A: DB Period (Up to Week 12)
Arm/Group | SC Placebo | IV Placebo | SC SAR441344 300 mg | IV SAR441344 1200 mg
Started | 14 | 12 | 51 | 52
Completed | 14 | 12 | 49 | 50
Not Completed | 0 | 0 | 2 | 2
Not completed — Adverse event: Related to Coronavirus Disease 2019 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Emergency situation due to war in Ukraine | 0 | 0 | 0 | 2
Period: Part B: OLE Period (Up to Week 296)
Arm/Group | SC Placebo | IV Placebo | SC SAR441344 300 mg | IV SAR441344 1200 mg
Started (After completing Part A, all participants entered Part B (OLE period), where participants in the IV and SC placebo arms switched to corresponding IV and SC SAR441344 arms) | 0 | 0 | 63 | 62
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 63 | 62
Not completed — Ongoing at the time of PCD | 0 | 0 | 63 | 62

BASELINE CHARACTERISTICS:
Population: The randomized population included all participants from screened population who were allocated to a randomized study drug by interactive response technology regardless of whether the study drug was received.
Groups:
- SC Placebo: Participants received placebo matched to SAR441344 IV infusion loading dose on Day 1 followed by placebo matched to SAR441344 SC injection on Weeks 2, 4, 6, 8 and 10 in Part A (DB period). At Week 12, all participants from this arm switched to active SC SAR441344 300 mg q2w and then switched to high SC SAR441344 dose of 1800 mg q4w in Part B (OLE period).
- Total: Total of all reporting groups
Arm/Group | SC Placebo | IV Placebo | SC SAR441344 300 mg | IV SAR441344 1200 mg | Total
Number analyzed (Participants) | 14 | 12 | 51 | 52 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.6 (10.8) | 32.3 (7.7) | 38.2 (8.9) | 37.3 (9.3) | 36.6 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 31 | 37 | 85
  Male | 4 | 5 | 20 | 15 | 44
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 0 | 0 | 1 | 0 | 1
  White | 14 | 12 | 50 | 52 | 128

OUTCOME MEASURES:

1. Primary Outcome: Mean Number of New Gadolinium (Gd)-Enhancing T1--Hyperintense (GdE T1) Lesions at Week 12 Relative to Week 8 as Measured by Brain Magnetic Resonance Imaging (MRI)
Description: Cranial (brain) MRI was performed to identify number of new GdE T1-hyperintense lesions at Week 12 relative to Week 8 MRI. Central review was used to identify new GdE T1 lesions not present at the previous MRI scans.
Time Frame: Week 8 and Week 12
Population: The efficacy population included all participants from the randomized population who took all Part A doses of study drug (1 SC dose skipped was allowed) and with an evaluable primary endpoint. As pre-specified in the statistical analysis plan (SAP), data for placebo arm is presented by pooling SC and IV placebo arms.
Measure: Least Squares Mean (95% Confidence Interval); unit: number of new GdE T1 lesions per month
Groups:
- Placebo: All participants received placebo matched to SAR441344 in Part A (DB period). At Week 12, all participants from this arm switched to active SAR441344 in Part B (OLE period).
Arm/Group | Placebo | SC SAR441344 300 mg | IV SAR441344 1200 mg
Number analyzed (Participants) | 22 | 45 | 47
number of new GdE T1 lesions per month | 1.4 [0.62 to 2.98] | 0.3 [0.13 to 0.59] | 0.2 [0.06 to 0.39]
Statistical Analysis 1: Comparison: Placebo vs SC SAR441344 300 mg; Negative binomial regression model adjusting for the categorical baseline GdE T1 lesion count (presence/absence) as covariate, treatment as factor, with offset equal to the log of the duration (in months) between the Week 12 MRI and previous MRI at Week 8; Test type: Superiority; Rate ratio = 0.21, 95% CI 2-sided [0.08 to 0.56]
Statistical Analysis 2: Comparison: Placebo vs IV SAR441344 1200 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Rate ratio = 0.11, 95% CI 2-sided [0.03 to 0.38]

2. Secondary Outcome: Mean Number of New or Enlarging T2 Lesions at Week 12 Relative to Week 8
Description: Cranial (brain) MRI was performed to identify number of new or enlarging T2 lesions at Week 12 relative to Week 8.
Time Frame: Week 8 and Week 12
Population: The efficacy population included all participants from the randomized population who took all Part A doses of study drug (1 SC dose skipped was allowed) and with an evaluable primary endpoint. As pre-specified in the SAP, data for placebo arm is presented by pooling SC and IV placebo arms.
Measure: Mean (Standard Deviation); unit: number of new or enlarging T2 lesions
Arm/Group | Placebo | SC SAR441344 300 mg | IV SAR441344 1200 mg
Number analyzed (Participants) | 22 | 45 | 47
number of new or enlarging T2 lesions | 3.8 (6.2) | 0.6 (1.8) | 0.3 (0.7)

3. Secondary Outcome: Mean Total Number of GdE T1 Lesions at Week 12
Description: Cranial (brain) MRI was performed to identify total number of GdE T1 lesions at Week 12.
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: number of GdE T1 lesions
Arm/Group | Placebo | SC SAR441344 300 mg | IV SAR441344 1200 mg
Number analyzed (Participants) | 22 | 45 | 47
number of GdE T1 lesions | 3.7 (7.4) | 0.5 (1.5) | 0.2 (0.5)

4. Secondary Outcome: Double-Blind Period: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: An AE was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study drug, whether or not considered related to the study drug. An SAE was any untoward medical occurrence that, at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect or was an important medical event. TEAEs were defined as AEs that developed, worsened or became serious during the TE period.
Time Frame: From first dose of study drug (Day 1) up to 12 weeks (DB TE period)
Population: The safety population included all randomized participants who took at least 1 dose (regardless of the amount) of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | SC Placebo | IV Placebo | SC SAR441344 300 mg | IV SAR441344 1200 mg
Number analyzed (Participants) | 14 | 12 | 51 | 52
Participants
  TEAEs | 5 | 3 | 23 | 15
  TESAEs | 0 | 0 | 0 | 0

5. Secondary Outcome: Double-Blind Period: Number of Participant With Anti-Drug Antibodies (ADAs) Against SAR441344
Description: Blood samples were collected at specified timepoints to assess the presence of ADAs against SAR441344. Treatment-emergent ADA was defined as at least 1 treatment-induced/boosted ADA. Treatment-induced ADA was defined as ADA that developed during the TE period and without pre-existing ADA (including participants without pre-treatment samples). Treatment-boosted ADA was defined as pre-existing ADA that was boosted during the TE period to a significant higher titer than the baseline. Number of participants with treatment-emergent ADA are presented.
Time Frame: From first dose of study drug (Day 1) up to 12 weeks (DB TE period)
Population: The ADA population included all participants from the safety population treated with SAR441344 in Part A with at least 1 post-baseline ADA result (positive, negative or inconclusive).
Measure: Count of Participants; unit: Participants
Arm/Group | SC Placebo | IV Placebo | SC SAR441344 300 mg | IV SAR441344 1200 mg
Number analyzed (Participants) | 14 | 12 | 51 | 51
Participants | 0 | 0 | 3 | 0

6. Secondary Outcome: Maximum Plasma Concentration (Cmax) of SAR441344
Description: Blood samples were collected at the specified timepoints for the assessment of Cmax. Cmax was assessed by a Bayesian approach using the population pharmacokinetic (PK) model.
Time Frame: After dose on Day 1 (first dose) and Weeks 8 (IV arm) and 10 (SC arm) (last dose)
Population: The PK population included all randomized and treated participants (safety population) with at least 1 post-baseline PK sample with adequate documentation of dosing and sampling dates and times. Only those participants with data collected at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: microgram per milliliter (mcg/mL)
Arm/Group | SC SAR441344 300 mg | IV SAR441344 1200 mg
Number analyzed (Participants) | 48 | 51
microgram per milliliter (mcg/mL)
  After first dose | 196 (34.4) | 623 (125)
  After last dose: number analyzed (Participants) | 46 | 50
  After last dose | 101 (20.9) | 580 (116)

7. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of SAR441344
Description: Blood samples were collected at the specified timepoints for the assessment of tmax. tmax was assessed by a Bayesian approach using the population PK model.
Time Frame: After dose on Day 1 (first dose) and Weeks 8 (IV arm) and 10 (SC arm) (last dose)
Population: The PK population included all randomized and treated participants (safety population) with at least 1 post-baseline PK sample with adequate documentation of dosing and sampling dates and times.
Measure: Median (Full Range); unit: hour
Arm/Group | SC SAR441344 300 mg | IV SAR441344 1200 mg
Number analyzed (Participants) | 48 | 51
hour
  After first dose | 1.5 [1 to 1.5] | 1.5 [1 to 2]
  After last dose: number analyzed (Participants) | 46 | 50
  After last dose | 97.2 [79 to 123] | 1.38 [0.92 to 1.77]

8. Secondary Outcome: Area Under the Curve Over the Dosing Interval (AUC0-tau) of SAR441344
Description: Blood samples were collected at the specified timepoints for the assessment of AUC0-tau. AUC0-tau was assessed by a Bayesian approach using the population PK model.
Time Frame: After dose on Day 1 (first dose) and Weeks 8 (IV arm) and 10 (SC arm) (last dose)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mcg*hour/mL
Arm/Group | SC SAR441344 300 mg | IV SAR441344 1200 mg
Number analyzed (Participants) | 48 | 51
mcg*hour/mL
  After first dose | 32800 (3560) | 157000 (23900)
  After last dose: number analyzed (Participants) | 46 | 50
  After last dose | 31900 (7580) | 190000 (39400)

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected from first dose of study drug (Day 1) up to 12 weeks (DB TE period). All-cause mortality (deaths) were collected from screening (Week -4) up to PCD of 21 September 2022, approximately up to 67 weeks
Description: Analysis was performed on safety population.
Arm/Group | SC Placebo | IV Placebo | SC SAR441344 300 mg | IV SAR441344 1200 mg
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/12 | 0/51 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/12 | 0/51 | 0/52
Other Adverse Events (participants affected / at risk) | 5/14 | 3/12 | 9/51 | 6/52
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SC Placebo (N=14) | IV Placebo (N=12) | SC SAR441344 300 mg (N=51) | IV SAR441344 1200 mg (N=52)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Hyperaemia (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Defaecation Urgency (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ingrowing Nail (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (3) | 0 (0)
Injection Site Erythema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection Site Extravasation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection Site Pain (General disorders) | 0 (0) | 1 (1) | 1 (4) | 1 (1)
Injury Associated With Device (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intentional Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2024-11-18): https://cdn.clinicaltrials.gov/large-docs/28/NCT04879628/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-18): https://cdn.clinicaltrials.gov/large-docs/28/NCT04879628/SAP_001.pdf